CLINICAL TRIAL: NCT01111552
Title: A Multicenter, Randomized, Double-blind Study to Evaluate the Efficacy, Safety and Tolerability of an Oral Aripiprazole/Escitalopram Combination Therapy in Patients With Major Depressive Disorder
Brief Title: Study to Evaluate the Efficacy, Safety and Tolerability of an Oral Aripiprazole/Escitalopram Combination Therapy in Participants With Major Depressive Disorder (MDD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early due to Sponsor decision, closure of this combination therapy program is unrelated to any safety issues, no signals of concern.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 31-08-256; 2010-018858-12 (EudraCT Number)
Record Dates: First submitted 2010-04-22; First posted 2010-04-27 (Estimated); Results first posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-09

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Major Depressive Disorder; MDD; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram; Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase B: Single-blind Prospective Treatment Phase (Active Comparator): Escitalopram 10 mg capsule, orally, once daily increased to 20 mg/day at the end of Week 1 based upon tolerability profile, plus one matching placebo capsule, for 8 weeks. No dose reductions were allowed after Week 4 and no dose increments were allowed after Week 3. Participants with incomplete response at the end of the Phase B (Week 8) entered Phase C and the rest of the participants continued to Phase B+.
  Interventions: Drug: Escitalopram; Drug: Placebo
- Phase B+: Single-blind Phase B Responders (Active Comparator): Participants with response at the end of the Phase B (Week 8) continued treatment with the single-blind escitalopram monotherapy at the dose (10 or 20 mg/day) taken during the final week of Phase B plus one matching placebo capsule, for an additional 6 weeks, in Phase B+.
  Interventions: Drug: Escitalopram; Drug: Placebo
- Phase C: Escitalopram Monotherapy (Active Comparator): Participants with incomplete response at Week 8 who were randomized to this arm group received escitalopram monotherapy 10 or 20 mg capsule, orally, once daily, whichever dose was taken during the final week of Phase B plus one matching placebo capsule for 6 weeks, in Phase C. No dose adjustments were allowed for escitalopram monotherapy during Phase C.
  Interventions: Drug: Escitalopram; Drug: Placebo
- Phase C: Aripiprazole Monotherapy (Active Comparator): Participants with incomplete response at Week 8 who were randomized to this arm group received aripiprazole 3, 6, or 12 mg capsule, orally, once daily plus one matching placebo capsule for 6 weeks, in Phase C. Participants were titrated to the aripiprazole target dose of 12 mg/day at Week 9 if the initial 6 mg/day dose was tolerated. No dose increments were allowed after Week 12; however, doses may have been decreased at any week, based upon tolerability.
  Interventions: Drug: Aripiprazole; Drug: Placebo
- Phase C: Aripiprazole/Escitalopram Combination Therapy (Active Comparator): Participants with incomplete response at Week 8 who were randomized to this arm group received aripiprazole 3, 6, or 12 mg capsule, orally, once daily in combination with the escitalopram 10 or 20 mg orally, once daily plus one matching placebo capsule for 6 weeks, in Phase C. No dose adjustments were allowed for escitalopram during Phase C. Participants were titrated to the aripiprazole target dose of 12 mg/day at Week 9 if the initial 6 mg/day dose was tolerated.
  Interventions: Drug: Escitalopram; Drug: Aripiprazole; Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — Escitalopram oral capsules.
  Arms: Phase B+: Single-blind Phase B Responders; Phase B: Single-blind Prospective Treatment Phase; Phase C: Aripiprazole/Escitalopram Combination Therapy; Phase C: Escitalopram Monotherapy
Drug: Aripiprazole — Aripiprazole oral capsules.
  Other Names: OPC-14597
  Arms: Phase C: Aripiprazole Monotherapy; Phase C: Aripiprazole/Escitalopram Combination Therapy
Drug: Placebo — Study drug matching placebo capsule.

SUMMARY:
This will be a multicenter, randomized, double-blind study designed to assess the efficacy, safety and tolerability of an oral Aripiprazole/Escitalopram combination therapy in participants with MDD who have demonstrated an incomplete response to a prospective trial of Escitalopram, and report a treatment history for the current MDD episode of an inadequate response to at least one and no more than three adequate trials of an approved antidepressant other than Escitalopram. An inadequate response is defined as less than a 50% reduction in depressive symptom severity as assessed by the participant's self-report on the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (ATRQ) and evaluated by the investigator as part of the participant's medical and psychiatric history. An adequate trial is defined as an antidepressant treatment for at least 6 weeks duration (or at least 3 weeks for combination treatments) at an approved dose as specified in the ATRQ.

DETAILED DESCRIPTION:
The study will be organized as follows:

* Screening Phase
* Single-blind Prospective Treatment Phase
* Single-blind Continuation Phase (Responder) or Double-blind Randomization Phase (non-Responder)
* 30 day Post Treatment Follow-up

Assigned Interventions:

* Escitalopram monotherapy
* Aripiprazole/Escitalopram combination therapy
* Aripiprazole monotherapy

ELIGIBILITY:
Inclusion Criteria:

* Participants with a current diagnosis of a major depressive episode. The current depressive episode must be ≥ 8 weeks in duration
* Participants willing to discontinue all prohibited psychotropic medication starting from the time of signing the informed consent and during the study period
* Participants with a 17-item Hamilton Depression Rating Scale (HAM-D17) total score ≥ 18 at the Baseline Visit for the Prospective Treatment Phase.

Exclusion Criteria:

* Lack of prior treatment with an antidepressant during the current depressive episode
* Participants who report treatment with adjunctive or monotherapy antipsychotic treatment during the current depressive episode.
* Participants experiencing hallucinations, delusions or any psychotic symptomatology in the current depressive episode
* Participants with epilepsy or significant history of seizure disorders
* Participants with a clinically significant current diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal or histrionic personality disorder
* Participants who have received electroconvulsive therapy (ECT) in the last 10 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2010-07-29 (Actual); Primary Completion 2011-09-27 (Actual); Study Completion 2011-09-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (54):
- United States (19):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Carson, California
  - Garden Grove, California
  - Imperial, California
  - Mission Viejo, California
  - Redlands, California
  - San Diego, California
  - Atlanta, Georgia
  - Hoffman Estates, Illinois
  - Terre Haute, Indiana
  - Overland Park, Kansas
  - Prairie Village, Kansas
  - Wichita, Kansas
  - Baltimore, Maryland
  - New York, New York
  - Toledo, Ohio
  - Bartlett, Tennessee
  - Wichita Falls, Texas
- Australia (5):
  - Brisbane, Queensland
  - Everton Park, Queensland
  - Malvern, Victoria
  - Melbourne, Victoria
  - Fremantle, Western Australia
- Bulgaria (10):
  - Burgas
  - Lovech
  - Novi Iskar
  - Pleven
  - Plovdiv
  - Rousse
  - Sofia
  - Tsarev Brod
  - Tserova Koria
  - Varna
- India (7):
  - Tirupati, Andhra Pradesh
  - Vijayawada, Andhra Pradesh
  - Manipal, Karnataka
  - Pune, Maharashtra
  - Ludhiana, Punjab
  - Chennai, Tamil Nadu
  - Kanpur, Uttar Pradesh
- Quezon City, NCR, Philippines
- Romania (7):
  - Bucharest
  - Study Site 1, Bucharest
  - Study Site 2, Bucharest
  - Craiova
  - Iași
  - Târgovişte
  - Târgu Mureş
- Slovakia (5):
  - Michalovce
  - Rimavská Sobota
  - Svidník
  - Trenčín
  - Zlaté Moravce

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 69 investigative sites in Australia, Bulgaria, India, Philippines, Romania, Russia, Slovakia, and the United States from 29 July 2010 to 27 September 2011.
Pre-assignment Details: A total of 237 major depressive disorder(MDD)participants were enrolled in Phase B(Single-blind Prospective Treatment Phase)to receive escitalopram monotherapy(10 or 20mg/day),of which 54 responders continued to Phase B+(Single-blind Phase B Responders),received escitalopram monotherapy(10 or 20mg/day).66 non-responders were randomized in 1:1:1 ratio to Phase C(Double-blind Randomization Phase),received escitalopram or aripiprazole monotherapy or aripiprazole/escitalopram combination therapy.
Period: Phase B (Day 1 to Week 8)
Arm/Group | Phase B: Single-blind Prospective Treatment Phase | Phase B+: Single-blind Phase B Responders | Phase C: Escitalopram Monotherapy | Phase C: Aripiprazole Monotherapy | Phase C: Aripiprazole/Escitalopram Combination Therapy
Started | 237 | 0 | 0 | 0 | 0
Completed | 120 | 0 | 0 | 0 | 0
Not Completed | 117 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 9 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0 | 0 | 0
Not completed — Sponsor Discontinued Study | 89 | 0 | 0 | 0 | 0
Not completed — Participant Met Withdrawal Criteria | 3 | 0 | 0 | 0 | 0
Not completed — Investigator Withdrew Participant | 3 | 0 | 0 | 0 | 0
Not completed — Participant Withdrew Consent | 7 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy as Determined by Investigator | 1 | 0 | 0 | 0 | 0
Period: Phase B+ and Phase C (Weeks 9 to 14)
Arm/Group | Phase B: Single-blind Prospective Treatment Phase | Phase B+: Single-blind Phase B Responders | Phase C: Escitalopram Monotherapy | Phase C: Aripiprazole Monotherapy | Phase C: Aripiprazole/Escitalopram Combination Therapy
Started | 0 | 54 | 22 | 21 | 23
Completed | 0 | 45 | 17 | 17 | 18
Not Completed | 0 | 9 | 5 | 4 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0
Not completed — Sponsor Discontinued Study | 0 | 5 | 4 | 3 | 5
Not completed — Participant Met Withdrawal Criteria | 0 | 2 | 0 | 0 | 0
Not completed — Investigator Withdrew Participant | 0 | 1 | 0 | 0 | 0
Not completed — Participant Withdrew Consent | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Phase B Sample included all participants who took at least one dose of escitalopram as indicated on the dosing record.
Arm/Group | Phase B: Single-blind Prospective Treatment Phase
Number analyzed (Participants) | 237
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156
  Male | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 218
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 30
  White | 186
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Phase C: Mean Change From End of Phase B (Week 8) in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score to End of Phase C (Week 14)
Description: The MADRS assessed severity of depressive symptoms. It ranges from a minimum of 0 to a maximum of 60 (higher scores indicating a greater severity of depressive symptoms). Participants are rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and a lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). A negative change from Week 8 indicates improvement. Last observation carried forward (LOCF) method was used for analyses.
Time Frame: Week 8 to Week 14
Population: Intent-to-treat (ITT) Sample included all participants in the Randomized Sample who received at least one dose of double-blind trial medication and had at least one post-randomization efficacy evaluation in Phase C.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase C: Escitalopram Monotherapy | Phase C: Aripiprazole Monotherapy | Phase C: Aripiprazole/Escitalopram Combination Therapy
Number analyzed (Participants) | 22 | 21 | 23
score on a scale | -8.0 (1.7) | -9.6 (1.7) | -9.2 (1.6)
Statistical Analysis 1: Comparison: Phase C: Escitalopram Monotherapy vs Phase C: Aripiprazole/Escitalopram Combination Therapy; Test type: Superiority; p = 0.595, ANCOVA; Treatment Difference = -1.3, 95% CI 2-sided [-5.9 to 3.4]
Statistical Analysis 2: Comparison: Phase C: Aripiprazole Monotherapy vs Phase C: Aripiprazole/Escitalopram Combination Therapy; Test type: Superiority; p = 0.869, ANCOVA; Treatment Difference = 0.4, 95% CI 2-sided [-4.4 to 5.1]

2. Secondary Outcome: Phase C: Clinical Global Impression - Improvement Scale (CGI-I) Score at The End of Phase C (Week 14)
Description: The CGI-I is a 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse. Last observation carried forward (LOCF) method was used for analyses.
Time Frame: Week 14
Population: ITT Sample included all participants in the Randomized Sample who received at least one dose of double-blind trial medication and had at least one post-randomization efficacy evaluation in Phase C.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Phase C: Escitalopram Monotherapy | Phase C: Aripiprazole Monotherapy | Phase C: Aripiprazole/Escitalopram Combination Therapy
Number analyzed (Participants) | 22 | 21 | 23
score on a scale | 2.4 (0.3) | 2.3 (0.2) | 2.3 (0.2)
Statistical Analysis 1: Comparison: Phase C: Escitalopram Monotherapy vs Phase C: Aripiprazole/Escitalopram Combination Therapy; Test type: Superiority; p = 0.856, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel Row Mean Scores Test was used to determine the p-value; Treatment Difference = -0.1, 95% CI 2-sided [-0.7 to 0.6]
Statistical Analysis 2: Comparison: Phase C: Aripiprazole Monotherapy vs Phase C: Aripiprazole/Escitalopram Combination Therapy; Test type: Superiority; p = 0.838, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel Row Mean Scores Test was used to determine the p-value; Treatment Difference = 0.1, 95% CI 2-sided [-0.6 to 0.7]

3. Secondary Outcome: Phase C: Mean Change From End of Phase B (Week 8) in the Sheehan Disability Scale (SDS) Mean Score to End of Phase C (Week 14)
Description: The SDS is a 3-item clinician-rated questionnaire used to evaluate impairments in the domains of work, social life/leisure, and family life/home responsibility. All items are rated on an 11-point continuum (0= no impairment to 10= most severe) with the total SDS score ranging from 0 (no impairment) to 30 (most severe). A negative change from Week 8 indicates improvement. Last observation carried forward (LOCF) method was used for analyses.
Time Frame: Week 8 to Week 14
Population: ITT Sample included all participants in the Randomized Sample who received at least one dose of double-blind trial medication and had at least one post-randomization efficacy evaluation in Phase C. Number analyzed is the number of participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase C: Escitalopram Monotherapy | Phase C: Aripiprazole Monotherapy | Phase C: Aripiprazole/Escitalopram Combination Therapy
Number analyzed (Participants) | 22 | 21 | 23
score on a scale | -0.9 (0.5) | -1.4 (0.5) | -1.2 (0.5)
Statistical Analysis 1: Comparison: Phase C: Escitalopram Monotherapy vs Phase C: Aripiprazole/Escitalopram Combination Therapy; Test type: Superiority; p = 0.765, ANCOVA; Treatment Difference = -0.2, 95% CI 2-sided [-1.6 to 1.2]
Statistical Analysis 2: Comparison: Phase C: Aripiprazole Monotherapy vs Phase C: Aripiprazole/Escitalopram Combination Therapy; Test type: Superiority; p = 0.760, ANCOVA; Treatment Difference = 0.2, 95% CI 2-sided [-1.2 to 1.6]

ADVERSE EVENTS:
Time Frame: From first dose of study drug through end of study (up to 22 weeks)
Description: Phase B Sample included all participants who took at least one dose of escitalopram as indicated on the dosing record. Phase B+ Sample included all participants who responded at the end of Phase B (were therefore not randomized) and who continued on single-blind escitalopram beyond Week 8. Randomized Sample included all participants who were randomized in Phase C.
Arm/Group | Phase B: Single-blind Prospective Treatment Phase | Phase B+: Single-blind Phase B Responders | Phase C: Escitalopram Monotherapy | Phase C: Aripiprazole Monotherapy | Phase C: Aripiprazole/Escitalopram Combination Therapy
All-Cause Mortality (participants affected / at risk) | 0/237 | 0/54 | 0/22 | 0/21 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/237 | 1/54 | 1/22 | 0/21 | 0/23
Other Adverse Events (participants affected / at risk) | 53/237 | 7/54 | 5/22 | 10/21 | 11/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase B: Single-blind Prospective Treatment Phase (N=237) | Phase B+: Single-blind Phase B Responders (N=54) | Phase C: Escitalopram Monotherapy (N=22) | Phase C: Aripiprazole Monotherapy (N=21) | Phase C: Aripiprazole/Escitalopram Combination Therapy (N=23)
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Physical assault (Social circumstances) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase B: Single-blind Prospective Treatment Phase (N=237) | Phase B+: Single-blind Phase B Responders (N=54) | Phase C: Escitalopram Monotherapy (N=22) | Phase C: Aripiprazole Monotherapy (N=21) | Phase C: Aripiprazole/Escitalopram Combination Therapy (N=23)
Nausea (Gastrointestinal disorders) | 18 | 0 | 2 | 1 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 1 | 0 | 2 | 2
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 2 | 2
Dizziness (Nervous system disorders) | 8 | 0 | 1 | 4 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 10 | 2 | 0 | 3 | 0
Weight increased (Investigations) | 2 | 2 | 0 | 0 | 2
Headache (Nervous system disorders) | 20 | 2 | 1 | 0 | 2
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to Sponsor decision, closure of this combination therapy program is unrelated to any safety issues, no signals of concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.